CLINICAL TRIAL: NCT00401791
Title: "ACTIV"Validation of a Paradigm for the Evaluation of Compounds That Activate Mitochondrial Biogenesis in Skeletal Muscle
Brief Title: ACTIV- Exercise Intervention in Healthy Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 26029
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2016-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Exercise
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — * Interval Exercise Training: Each interval training session will start with 10 minutes of warm up and will end with 10 minutes of cool down period at 40% VO2 peak. Training duration, intensity and number of exercise bout will increase with the progression of training period
  * Aerobic training: Each endurance training session will start with 5 minutes of warm up and will end with 5 minutes of cool down at 40% VO2 peak. Subjects will exercise at 70% VO2 peak for 45 minutes on day 3 and 5, for 55 minutes on day 8 and 10, and for 35 minutes on day 14 using a bicycle ergometer.
  Other Names: Aerobic and interval exercise training
  Arms: 1

SUMMARY:
The study is designed to compare muscle energy capacity in men with obesity or diabetes as compared to athletes. This study will also enable researchers to determine whether MRS can replace muscle biopsy for this type of assessment.

DETAILED DESCRIPTION:
Skeletal muscle mitochondrial defects are a sine qua non of insulin resistance in patients with type 2 diabetes mellitus (T2DM), obese and subjects with family history of T2DM (FH+). Exercise increases mitochondrial capacity whereas lipid infusion or high fat diet decreases genes involved in mitochondrial biogenesis. In this study 2 cohorts will be involved: Cohort I (athletes, T2DM and obese) and Cohort II (healthy with "FH+" or without "FH-" family history of T2DM). This randomized, parallel arm clinical trial will consist of 4 periods: screening, stabilization (3 days), baseline (for Cohort I and II) and exercise period (14 days, only for Cohort II). The overall objective of the study is to validate a paradigm for the evaluation of compounds and drugs that activate mitochondrial biogenesis in skeletal muscle. In Specific Aim 1 we will compare and contrast biopsy and MRS power to detect differences in mitochondrial capacity in 78 subjects: athletes (N=10), FH- (N=24), FH+ (N=24), obese (N=10) and T2DM (N=10). In Specific Aim 2 we will compare mitochondrial changes in response to exercise in subjects FH - vs. FH + subjects. In Specific Aim 3 we will determine if HFD impairs mitochondrial changes in response to exercise in FH+ subjects. In Specific Aim 4 we will determine the role of mitochondrial capacity in metabolic flexibility and insulin sensitivity in T2DM, obese, FH+, FH- and athlete subjects.

ELIGIBILITY:
Inclusion Criteria:

T2DM group:

* Men aged 25-35
* BMI > 30 kg/m2
* Sedentary lifestyle determined by activity index questionnaire (not involved in regular exercise program) and accelerometer data.
* Are willing to eat only foods provided by Pennington for the study period
* Diagnosed with T2DM defined by one or more of the following:

  * fasting plasma glucose > 126 mg/dL at entry
  * a two-hour OGTT glucose > 200mg/dL
  * current medication for T2DM

Obese group:

* Men aged 25-35
* BMI > 30 kg/m2
* Sedentary lifestyle activity index questionnaire (not involved in regular exercise program) and accelerometer data.
* Are willing to eat only foods provided by Pennington for the study period

FH+ group:

* Men aged 25-35
* One parent diagnosed with T2DM
* fasting insulin > 10mIU/ml (> 50th %tile)
* BMI between 22 and 30 kg/m2
* Sedentary lifestyle activity index questionnaire (not involved in regular exercise program) and accelerometer data.
* Are willing to exercise every day for the study period
* Are willing to eat only foods provided by Pennington for the study period

FH- group:

* Men aged 25-35
* Parents and grandparents were not diagnosed with T2DM
* Fasting insulin < 10mIU/ml (< 50th %tile)
* BMI between 22 and 30 kg/m2
* Sedentary lifestyle activity index questionnaire (not involved in regular exercise program) and accelerometer data.
* Are willing to exercise for the study period
* Are willing to eat only foods provided by Pennington for the study period

Athlete group:

* Men aged 25-35
* Maximal oxygen uptake > 60 ml/kg.min
* Are engaged in minimum of 1.5 h of aerobic exercise 3 times/ week
* Are willing to eat only foods provided by Pennington for the study period

Exclusion Criteria:

* Abnormal resting or exercise ECG
* Significant renal, cardiac, liver, lung, or neurological disease (controlled hypertension is acceptable if baseline bp < 140/90 on medications)
* Use of drugs known to affect energy metabolism or body weight: including, but not limited to: orlistat, sibutramine, ephedrine, phenylpropanolamine, corticosterone, etc
* Alcohol or other drug abuse
* Smoking
* Gait problems
* Unwilling or unable to abstain from caffeine (48h) prior to metabolic rate measurements
* Unwilling or unable to eat all study foods
* Increased liver function tests at baseline (AST/ALT/GGT/or alkaline phosphatase greater than 2.5 times the upper limit of normal)
* Metal objects that would interfere with the measurement of body composition /MRS such as implanted rods, surgical clips, etc
* NYHA class III/IV CHF is an exclusionary cardiac condition
* history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* varicose veins
* major surgery on the abdomen, pelvis, or lower extremities within previous 3 months
* cancer (active malignancy with or without concurrent chemotherapy)
* rheumatoid disease
* bypass graft in limb
* known genetic factor (Factor V Leiden, etc) or hypercoagulable state
* diagnosed peripheral arterial or vascular disease, or intermittent claudication
* family history of primary DVT or PE (pulmonary embolism)
* peripheral neuropathy

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To compare/ contrast the power of skeletal muscle biopsy vs. MRS to detect differences in mitochondrial capacity | baseline and after intervention

SECONDARY OUTCOMES:
To compare mitochondrial changes in response to exercise in subjects FH - vs. FH + subjects by skeletal muscle biopsy and MRS | baseline and after intervention
To determine if HFD impairs mitochondrial changes in response to exercise in the FH + group by muscle biopsy and MRS. | baseline and after intervention
To determine the role of mitochondrial capacity in metabolic flexibility and insulin sensitivity | baseline and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Covington JD, Noland RC, Hebert RC, Masinter BS, Smith SR, Rustan AC, Ravussin E, Bajpeyi S. Perilipin 3 Differentially Regulates Skeletal Muscle Lipid Oxidation in Active, Sedentary, and Type 2 Diabetic Males. J Clin Endocrinol Metab. 2015 Oct;100(10):3683-92. doi: 10.1210/JC.2014-4125. Epub 2015 Jul 14. PMID 26171795
- [Derived] Bajpeyi S, Myrland CK, Covington JD, Obanda D, Cefalu WT, Smith SR, Rustan AC, Ravussin E. Lipid in skeletal muscle myotubes is associated to the donors' insulin sensitivity and physical activity phenotypes. Obesity (Silver Spring). 2014 Feb;22(2):426-34. doi: 10.1002/oby.20556. Epub 2013 Sep 10. PMID 23818429
- [Derived] Gan Z, Rumsey J, Hazen BC, Lai L, Leone TC, Vega RB, Xie H, Conley KE, Auwerx J, Smith SR, Olson EN, Kralli A, Kelly DP. Nuclear receptor/microRNA circuitry links muscle fiber type to energy metabolism. J Clin Invest. 2013 Jun;123(6):2564-75. doi: 10.1172/JCI67652. Epub 2013 May 8. PMID 23676496
- [Derived] Bajpeyi S, Pasarica M, Moro C, Conley K, Jubrias S, Sereda O, Burk DH, Zhang Z, Gupta A, Kjems L, Smith SR. Skeletal muscle mitochondrial capacity and insulin resistance in type 2 diabetes. J Clin Endocrinol Metab. 2011 Apr;96(4):1160-8. doi: 10.1210/jc.2010-1621. Epub 2011 Feb 9. PMID 21307136
- [Derived] Costford SR, Bajpeyi S, Pasarica M, Albarado DC, Thomas SC, Xie H, Church TS, Jubrias SA, Conley KE, Smith SR. Skeletal muscle NAMPT is induced by exercise in humans. Am J Physiol Endocrinol Metab. 2010 Jan;298(1):E117-26. doi: 10.1152/ajpendo.00318.2009. Epub 2009 Nov 3. PMID 19887595